CLINICAL TRIAL: NCT04580901
Title: Out-patient Group Therapy Using Interpersonal Psychotherapy for Mums With Postpartum Depression: the OPTIMUM Study: a Randomized Controlled Trial
Brief Title: IPT-G for Mums With Postpartum Depression
Acronym: OPTIMUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Hamilton Academic Health Sciences Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10612
Record Dates: First submitted 2020-09-25; First posted 2020-10-09 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Postpartum Depression
Keywords: postpartum; perinatal; depression; depressive disorder
MeSH Terms: conditions — Depression, Postpartum; Depression; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group interpersonal psychotherapy (Experimental): Group IPT consists of 12 weeks of virtually delivered therapy by two co-therapists via Zoom to a group of 6-8 women. The 12 weeks consist of 15 sessions over 12 weeks of group IPT taking place virtually via Zoom (2 sessions per week for the first 4 weeks (acute phase) then once a week for 6 weeks, then a two-week space before the last session).
  Interventions: Behavioral: Group Interpersonal Psychotherapy
- Usual care (No Intervention): Usual care refers to any care that the women wish to access, and there are no limits on the women in either group. It may include, but is not limited to, the family physician, obstetrician, and/or midwife, participation in regional standard perinatal depression programming, private therapy, online therapies, medication, etc.

INTERVENTIONS:
Behavioral: Group Interpersonal Psychotherapy — Group IPT consists of 12 weeks of virtually delivered therapy by two co-therapists via Zoom to a group of 6-8 women. The 12 weeks consist of 15 sessions over 12 weeks of group IPT taking place virtually via Zoom (2 sessions per week for the first 4 weeks (acute phase) then once a week for 6 weeks, then a two-week space before the last session).
  Other Names: Group IPT
  Arms: Group interpersonal psychotherapy

SUMMARY:
Postpartum depression is a very common and costly illness with numerous, long-term deleterious effects for women, their offspring and families; yet most women are not treated. Group IPT delivered virtually offers women a 1st-line, low-cost intervention that overcomes existing treatment barriers. To test its acceptability and effectiveness, a RCT will be conducted to compare virtually delivered group IPT immediately to usual care in women in Ontario Canada who have postpartum depression.

DETAILED DESCRIPTION:
Depression during pregnancy and in the first year following delivery affects 15-20% of women. Left untreated, these disorders increase the risk of future depressive episodes, postpartum depression in their partners, as well as emotional, behavioural, and cognitive problems in offspring. Unfortunately, up to 85% of these women will not receive treatment, which is estimated to cost the province of Ontario upwards of $6 billion annually. There is significant stigma surrounding perinatal depression which can result in less help-seeking by women, as well as a lack of awareness about available non-medication treatment options among both physicians and patients, even though most women prefer psychotherapy over medication.

Despite the very strong evidence base for IPT, relatively few clinicians are trained to deliver IPT. Rather than travelling to tertiary care centres, the delivery of group psychotherapy virtually via telemedicine or Zoom allows women anywhere in the province to access this highly effective first-line treatment, thereby increasing access for women with perinatal depression and improving outcomes for mothers, babies, and families in Ontario.

Study Objective: To compare the effectiveness of virtual group IPT to usual care in women with postpartum depression symptoms for reducing depression symptoms and anxiety, improving mother-infant attachment, and increasing social support, functioning, and quality of life.

Study Design: RCT Population: postpartum women, aged 18 or older, with a baby under a year old Intervention: 12 weeks (15 sessions - 12 acute, 3 maintenance sessions) of group IPT delivered virtually via Zoom Comparison: 12 weeks of usual care followed by group IPT Outcomes: Pre-treatment versus post-treatment change in depression symptoms, anxiety, acceptability, mother-infant bonding, social support & functioning, and quality of life.

All women in the study will be able to access care as usual from their physicians and other therapists throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* postpartum with baby under 1 year
* score greater than or equal to 10 on the Edinburgh Postnatal Depression Scale (EPDS)

Exclusion Criteria:

* active alcohol or substance use disorder
* bipolar disorder
* borderline personality
* antisocial personality
* PTSD
* psychosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 95 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms on Edinburgh Postpartum Depression scale | To be measured immediately after 12 weeks of group IPT
  Pre-treatment to post-treatment comparison of depressive symptoms measured via EPDS. Scale is measured from 1 (no depressive symptoms) to 4 (worst depressive symptoms) with 0 being the lowest score (best outcome) and 30 being the highest score (worst outcome).
Depressive symptoms on Patient Health Questionnaire-9 (PHQ-9) | To be measured immediately after 12 weeks of group IPT
  Pre-treatment to post-treatment comparison of depressive symptoms measured via PHQ-9. Scale is measured from 0 (no depressive symptoms) to 3 (worst depressive symptoms) with 0 being the lowest score (best outcome) and 27 being the highest score (worst outcome).

SECONDARY OUTCOMES:
Anxiety | Immediately after 12 weeks of group IPT
  Pre-treatment to post-treatment comparison of anxiety symptoms measured via Generalized Anxiety Disorder-7 scale. Scale is measured from 0 (least anxiety) to 3 (most anxiety) with 0 being the lowest score (best outcome) and 21 being the highest score (worst outcome).
Acceptability | Immediately after 12 weeks of group IPT
  Acceptability of the treatment as measured by Client Satisfaction Questionnaire-8. Scale is measured from 1 (least satisfied) to 4 (most satisfied) with 8 being the lowest score (worst outcome) and 32 being the highest score (best outcome).
Social Support | Immediately after 12 weeks of group IPT
  Pre-treatment to post-treatment comparison of social supports using the Social Provisions Scale. This 24-item scale is measured from 1 (strongly disagree) to 4 (strongly agree) with 24 being the lowest score (worst outcome) and 96 being the highest score (best outcome).
Functioning | Immediately after 12 weeks of group IPT
  Pre-treatment to post-treatment comparison of functioning using the Sheehan Disability Scale. Scale is measured from 0 (not at all disrupted) to 10 (extremely disrupted) with 0 being the lowest score (best outcome) and 30 being the highest score (worst outcome).
Anxiety | Immediately after 12 weeks of group IPT
  Pre-treatment to post-treatment comparison of anxiety symptoms measured via Zung Self-Rating Anxiety scale. Scale is measured from 1 (least anxiety) to 4 (most anxiety) with 20 being the lowest score (best outcome) and 80 being the highest score (worst outcome).
Postpartum bonding | Immediately after 12 weeks of group IPT
  Postpartum Bonding Questionnaire will be used to measure maternal-infant attachment pre- and post-treatment. This 25-item scale is measured from 0 (least bonded) to 5 (most bonded) with 0 being the lowest score (worst outcome) and 125 being the highest score (best outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Polak, HBA BMSc MD, Principal Investigator — McMaster University
Locations (1):
- McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No